CLINICAL TRIAL: NCT03047473
Title: Avelumab in Patients With Newly Diagnosed Glioblastoma Multiforme
Acronym: SEJ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinique Neuro-Outaouais (Other)
Responsible Party: Principal Investigator, Dr. Francois Jacques, neurologist, Clinique Neuro-Outaouais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNO-006
Record Dates: First submitted 2017-01-31; First posted 2017-02-09 (Estimated); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: newly diagnosed
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Intervention Model Description: single center, add on, open label, single dose, single arm
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Newly diagnosed GBM (Experimental): single arm, open label Addition of Avelumab to standard treatment
  Interventions: Biological: avelumab

INTERVENTIONS:
Biological: avelumab — add on of avelumab 10mg/kg IV to standard therapy

SUMMARY:
This is a safety and tolerability study looking at the addition of avelumab, an immune checkpoint inhibitor, to standard therapy of temozolomide and radiotherapy in patients with newly diagnosed glioblastoma multiforme.

All patients will be receiving active therapy. Patients will begin the avelumab within 3 weeks of finishing their radiotherapy. Avelumab will be given at a dose of 10mg/kg IV every 2 weeks concomitantly with the monthly temozolomide. Avelumab will be continued for a total of 52 weeks.

DETAILED DESCRIPTION:
Protocol Title: Avelumab in patients with newly diagnosed Glioblastoma Multiforme

Indication: Patients with newly diagnosed Glioblastoma Multiforme

Study Type: Single center, phase 2, open ended, open label addition of avelumab to standard therapy

Objectives

Primary Objectives:

To determine the safety and tolerability of avelumab administered as 10mg/kg IV q2weeks in patients receiving standard therapy for newly diagnosed GBM.

Secondary objectives:

To determine the impact of the addition of avelumab at a dose of 10mg/kg IV Q2weeks in patients receiving standard therapy for newly diagnosed GBM on overall survival (OS), progression free survival (PFS) and other antitumor activity parameters according to the immunotherapy Response Assessment for Neuro-Oncology (iRANO) (1) at 52 weeks.

Exploratory objectives:

To explore biomarkers that could predict treatment response to avelumab such as: the tumor immunoscore, presence and extent of PD-L1 expression on tumor cells and microglia/macrophages within the tumor

To correlate the OS and PFS in relation to the change between baseline and end of study neurocognitive function as measured by the evoked potential P300 (normal), the baseline corticosteroid dose, the average daily corticosteroid dose over the whole study duration, those who for tolerability reasons do not complete the temozolomide standard 6 monthly pulses of therapy and the presence and severity of immune related adverse events (irAE's).

To assess and compare above mentioned biomarkers in tissue samples from patients with second surgical resection ie treatment failures.

To assess in this GBM population the duration of pseudoprogression and the lagtime needed for immunotherapy to become effective.

Study Design: This is a single center, phase 2, open label, add-on, single dose study in patients receiving standard therapy for newly diagnosed GBM. In total 30 patients who meet the entry criteria will be entered into the study within 3 weeks of finishing their last day of combined radiotherapy/temozolamide. Avelumab will be initiated concurrently with the initiation of the first 5 day, monthly cycle of temozolamide and continued for a total of 260 weeks.

A local pathology report will constitute adequate documentation of histology for study inclusion.

The tumor block used for diagnosis of GBM must be collected for each patient and sent for MGMT assessment (if not already done), biomarker and immunoscore analysis. The availability of these samples is mandatory for randomization into the study, and they must be sent within 2 months after patient's entry into the study for analysis.

Paraffin embedded blocks containing formalin-fixed tumor tissue representative of the glioblastoma diagnosis is the preferred sample (if available, and of sufficient quality), otherwise, a partial tumor block, or pathology material should be sent. If surgery was not performed but biopsy was performed (or if it is not possible to send FFPE tumor tissue blocks) at least 10 unstained, uncovered slides must be sent.

The study will consist of 3 different phases: a Combination Phase, a Monotherapy Phase and an Extended Safety Follow-up Phase

Combination Phase: Upon completion of the standard combination therapy of radiotherapy (total dose 60 Gy, administered as daily 2Gy fractions, 5 days/week) and temozolomide (75 mg/m2/day p.o. qd) and a treatment break of no more than 21 days, the combination phase will start. Patients will receive temozolomide and avelumab for 6 cycles of 28 days each. During the 1st cycle Temozolomide will be given the first 5 days at a dose of 150mg/m2/day p.o. In the next cycle, the temozolomide dose should be escalated to 200/mg/m2 if permitted by the patient's hematological and non-hematological toxicity profile (as per NCI-CTC AE version 3). The temozolomide dose will be adjusted according to hematological and non-hematological toxicity as per temozolomide's product monograph (appendix 4). Avelumab will be administered on day 1 and day 15 of each cycle at a dose of 10mg/kg IV. Avelumab therapy will be withheld according to the occurrence and severity of avelumab related adverse events as per table 3. Patients will continue the combination of temozolomide (150-200mg/m2 per day PO X5 days Q28days) and avelumab (at 10mg/kg dose, IV on days 1 and 15 per cycle) until 6 cycles are completed or until confirmed disease progression or unacceptable (grade 3 or higher) avelumab related toxicity occurs.

Monotherapy Phase: Upon completion of the Combination Phase or upon stopping temozolomide because of temozolomide related toxicity the patient will continue into the avelumab Monotherapy Phase. Avelumab 10mg/kg IV Q2weeks will be continued as monotherapy until a total of 260 weeks of avelumab has been received or evidence of confirmed disease progression as per the iRANO definition or unacceptable (grade 3 or higher) avelumab related toxicity has occurred.

Patients who experience irAE's may according to table 3 directives have their avelumab therapy suspended.

The use of Bevacizumab, second surgical resection or re-irradiation will not be allowed in the study and will be considered as evidence of disease progression.

Patients will be promptly informed upon confirmation of disease progression as per the new iRANO criteria. They will be offered to pursue with the avelumab therapy as per protocol or to withdraw from therapy and enter the extended safety follow up phase.

Upon completion of the Monotherapy Phase at week 260 patients will be then be offered the option of being rolled over into an open label extension study or receive commercial avelumab via a special access program.

Extended Safety Follow-up Phase:

Patients who discontinue avelumab therapy for any reason at any point in the study will be entered into an extended safety follow-up period of 90 days. Treatment will then be at the investigator or local oncologist's discretion. All subjects will be observed for the possible occurrence of delayed irAE's. Survival data and information about subsequent therapies will be collected. Tissue samples in patients undergoing second surgical resections will be obtained for further biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥ 18 years.
3. Present with newly diagnosed supratentorial Glioblastoma (GBM) with a tissue diagnosis that has been established following either a surgical resection or biopsy. This includes treatment-naïve -(chemotherapy and radiotherapy)- patients with prior diagnosis of a lower grade astrocytoma that has been upgraded to a histologically verified GBM.
4. Karnofsky performance score of 70 or higher.
5. Patients entering the study must be on a stable dose of up to 12 mg (maximum) of Dexamethasone (or equivalent) daily for symptoms related to cerebral edema. Following the first dose of avelumab, the duration of treatment with the current dose of dexamethasone (maximum 12 mg/day) or equivalent, should be no more than 7 consecutive days. The investigator(s) should make every effort to taper the dexamethasone as soon as symptom improvement allows to the lowest tolerable dose that controls the CNS symptoms.
6. Will be or is undergoing or has received the standard therapy of chemo radiation therapy (60Gy in 30 fractions of 2Gy/day with concurrent temozolomide of 75mg/m2 per day PO) no more than 21 days ago.
7. Has not yet begun but will begin standard monthly temozolomide therapy.
8. Patient must have at least 1 formalin fixed paraffin embedded tumor tissue block representative of glioblastoma available for biomarker analysis and determination of MGMT status (if not already done). If tumor block is not available or not of adequate quality, sufficient pathology material, representative of glioblastoma, must be available.
9. Adequate hematological function defined by absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused).
10. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN for all subjects.
11. Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
12. Negative serum pregnancy test at screening for women of childbearing potential.
13. Highly effective contraception for both male and female subjects if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1 % per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 60 days after avelumab treatment.
14. International normalized ratio (INR) or PT (secs) and activated partial thromboplastin time (aPTT):

    * in the absence of therapeutic intent to anticoagulate the subject: INR≤1.5 or PT ≤1.5 x ULN and aPTT ≤1.5 x ULN
    * in the presence of therapeutic intent to anticoagulate the subject: INR or PT and aPTT within therapeutic limits (according to the medical standard in the institution).

    NOTE: Use of full-dose anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to randomization.
15. Willing and able to comply with the protocol as judged by the Investigator

Exclusion Criteria:

1. Patients who have evidence of leptomeningeal disease.
2. Known significant pulmonary, cardiovascular, hepatic disorders or any other disease that in the opinion of the investigator would be contraindicated to receive anti PD-L1 therapy such as avelumab.
3. Prior treatment with bevacizumab or any checkpoint immune blockade thérapies.
4. Any other concomitant immunosuppressant other than temozolamide and steroids or any recent (within 3 months) experimental therapy.
5. Patients who have finished their radiotherapy course more than 3 weeks prior to Baseline.
6. Prior organ transplantation, including allogeneic stem cell transplantation.
7. Significant acute or chronic infections including, among others:

   * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
   * Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive).
8. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

   * Subjects with diabetes type I, vitiligo, psoriasis, hypo or hyperthyroid disease or any other autoimmune disease not requiring immunosuppressive treatment are at the investigator's discretion eligible
   * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
   * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable.
9. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
10. Pregnancy or lactation.
11. Known alcohol or drug abuse.
12. Any psychiatric or cognitive condition that would prohibit the understanding or rendering of informed consent.
13. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines.
14. Contraindication or intolerance to temozolomide.
15. Any other malignancy within 5 years prior to randomization, except for adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix.
16. Evidence of any active infection requiring hospitalization or IV antibiotics within 2 weeks prior to randomization.
17. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
18. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Jacques, MD, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada

REFERENCES:
- [Derived] Jacques FH, Nicholas G, Lorimer IAJ, Sikati Foko V, Prevost J, Dumais N, Milne K, Nelson BH, Woulfe J, Jansen G, Apedaile BE. Avelumab in newly diagnosed glioblastoma. Neurooncol Adv. 2021 Aug 25;3(1):vdab118. doi: 10.1093/noajnl/vdab118. eCollection 2021 Jan-Dec. PMID 34604752
- See also: GBM clinical trial website — https://www.gbmtherapy.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolment began 19 May 2017 and ended 04 August 2021 Enrollmenet was conducted at the study site : Clinique Neuro-Outaouais
Pre-assignment Details: 430 candidates were prescreened 38 were screened with 30 randomized The reasons for screen failure included: blood abnormality (n=3) withdrawal of consent (n=4) and low Karnofsky score (n=1)
Period: Overall Study
Arm/Group | Newly Diagnosed GBM
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Newly Diagnosed GBM
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 30
MGMT methylation status [Count of Participants; unit: Participants]
  MGMT methylated | 10
  MGMT unmethylated | 16
  MGMT status unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: The number of patients with an avelumab related adverse event leading to permanent or transient discontinuation of avelumab treatment.
  Treatment related adverse events of special interest will include those of autoimmune origin (irAE).
  The adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0
Time Frame: over the course of the 52 weeks stsudy
Measure: Number; unit: participants
Arm/Group | Newly Diagnosed GBM
Number analyzed (Participants) | 30
participants
  tumor progression | 19
  radiation necrosis | 2
  seizure | 2
  thrombotic event | 2
  liver enzymes elevation | 3
  other | 12

2. Secondary Outcome: Safety and Tolerability
Description: The number of Participants with an Emergent Adverse Event Leading to Avelumab Interruption or Termination
Time Frame: over the course of the 52 weeks study
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed GBM
Number analyzed (Participants) | 30
Participants | 3

ADVERSE EVENTS:
Time Frame: over the course of 52 weeks of the study
Arm/Group | Newly Diagnosed GBM
All-Cause Mortality (participants affected / at risk) | 26/30
Serious Adverse Events (participants affected / at risk) | 27/30
Other Adverse Events (participants affected / at risk) | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Newly Diagnosed GBM (N=30)
tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 (27) — secondary progression of their glioblastoma
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Newly Diagnosed GBM (N=30)
hepatic enzymes elevation (Hepatobiliary disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT03047473/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT03047473/SAP_002.pdf